CLINICAL TRIAL: NCT06493357
Title: UNCPM 22401 - Evaluation of a Differentiated Point-of-care Active Case Finding & Management Model for the Elimination of Mother-to-Child Transmission of HIV in Lilongwe and Mangochi, Malawi
Brief Title: Evaluation of a Differentiated Point-of-care Active Case Finding & Management Model to Eliminate Mother-to-Child Transmission of HIV in Malawi
Acronym: PAC-Man
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0561; 1P01HD112215 (NIH)
Record Dates: First submitted 2024-06-26; First posted 2024-07-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: HIV Prevention
Keywords: HIV Treatment
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAC-Man Model (Experimental): PAC-Man represents an integrated DSD model for mothers and infants that brings the following three evidence-based practices into the community for EMTCT: 1) pediatric active case finding using novel POC EID technology; 2) same-day ART initiation for infants newly diagnosed with HIV infection; and 3) mVL testing and back-to-care services. PAC-Man uses a mobile approach to offer EMTCT services in the community and reach "high risk" MIPs. Delivering the PAC-Man model will be done under the auspices of routine care, applying an overarching implementation strategy of creating new mobile care teams equipped with new diagnostic technology who deploy the m-PIMA in community settings.
  Interventions: Behavioral: PAC-Man
- Standard of care (control arm) (Active Comparator): Routine care as provided by the Ministry of Health.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: PAC-Man — PAC-Man represents an integrated DSD model for mothers and infants that brings the following three evidence-based practices into the community for EMTCT: 1) pediatric active case finding using novel POC EID technology; 2) same-day ART initiation for infants newly diagnosed with HIV infection; and 3) mVL testing and back-to-care services. PAC-Man uses a mobile approach to offer EMTCT services in the community and reach "high risk" MIPs. Delivering the PAC-Man model will be done under the auspices of routine care, applying an overarching implementation strategy of creating new mobile care teams equipped with new diagnostic technology who deploy the m-PIMA in community settings.
  Arms: PAC-Man Model
Behavioral: Standard of Care — Routine care as provided by Ministry of Health.
  Arms: Standard of care (control arm)

SUMMARY:
Purpose: To conduct a hybrid effectiveness-implementation stepped-wedge trial to:

1. Estimate the effect of the PAC-Man model, compared to SOC, on the proportion of infants who receive timely EID testing.
2. Estimate the effect of the PAC-Man model, compared to SOC, on the proportion of pregnant and breastfeeding women living with HIV who receive guideline-adherent viral load testing.
3. Compare implementation outcomes between the PAC-Man model and SOC.

Participants: The total study sample size is 2,426, including 2,304 mother-infant pair (MIP) survey participants, 48 high-risk pregnant/breastfeeding women living with HIV for in-depth interviews (from high-risk MIPs who participated in a survey); 10 PMTCT policy makers and Ministry of Health (MOH)/ President's Emergency Plan for AIDS Relief (PEPFAR) implementing partner senior managers for key informant interviews; and about 48-64 professional and lay health providers for focus group discussions and implementation actor surveys.

To rigorously evaluate the PAC-Man model, investigators will use a hybrid (type 3) effectiveness-implementation incomplete stepped-wedge trial design. The hybrid incomplete stepped-wedge design is a rigorous quasi-experimental design that allows for incremental "rollout" of the PAC-Man model and serial measurement of both health outcomes (for infants and mothers in Objectives 1 and 2, respectively), as well as implementation outcomes (Objective 3). The incomplete stepped-wedge design is more efficient than a complete design, minimizes costs, and reduces participant burden, without sacrificing statistical precision. Using this design, sequential crossover from control (i.e., the SOC) to intervention (i.e., SOC plus the PAC-Man model) takes place at each 'step' using cluster randomization until all clusters (defined as a group of "sites," or health facilities plus the surrounding communities in its catchment area) receive the intervention. The 12 sites included in our study will be divided into 4 clusters of 3 sites each.

DETAILED DESCRIPTION:
PAC-Man Model:

PAC-Man represents an integrated differentiated services delivery (DSD) model for mothers and infants that brings the following three evidence-based practices into the community for elimination of mother to child transmission (EMTCT): 1) pediatric active case finding using novel point-of-care (POC) early infant diagnosis (EID) technology; 2) same-day antiretroviral therapy (ART) initiation for infants newly diagnosed with HIV infection; and 3) maternal viral load (mVL) testing and back-to-care services. PAC-Man uses a mobile approach to offer EMTCT services in the community and reach "high risk" MIPs in which the mother living with HIV did not initiate ART, started ART late during pregnancy or breastfeeding, dropped off treatment following ART initiation, was unsuppressed on ART, was identified with HIV infection for the first-time during the post-partum period, and/or did not return with her infant for EID testing. Because these evidence-based practices are already recommended by the Ministry of Health and will be functioning at the site and not the individual level, delivering the PAC-Man model will be done under the auspices of routine care, applying an overarching implementation strategy of creating new mobile care teams equipped with new diagnostic technology who deploy the m-PIMA™ in community settings.

PAC-Man Implementation Approaches:

The overall implementation strategy being evaluated in this study is the creation of mobile care teams to deploy m-PIMA™ and provide EMTCT services in the community. Complementing this overarching strategy will be two sub-strategies used to enhance PAC-Man adoption: 1) task shifting of active case finding, EID and mVL testing, ART initiation, and back-to-care services to community health workers (CHWs), community nurses, and HIV diagnostic assistants; and 2) changing service sites to convenient locations in the community to overcome barriers to EID and mVL delivery. These strategies are intended to work in concert with the above evidence-based practices to integrate PAC-Man into the EMTCT program.

ELIGIBILITY:
The criteria for Enumerated MIP Cohort is as follows:

Inclusion Criteria:

* Enrolled in the national EMTCT program at a study site in the 12 months preceding a survey.

Exclusion Criteria:

* None.

The criteria for Enumerated MIP Field Survey is as follows:

Inclusion Criteria:

* Age 16 years or older.
* Enrolled in the national EMTCT program at a study site in the 12 months preceding a survey.

Exclusion Criteria:

* Documented transferred out from a site prior to the field survey.
* Participated previously in the field survey.
* Decline informed consent.

The criteria for In-Depth Interviews is as follows:

Inclusion criteria:

* Age 16 years or older.
* Met high-risk criteria for PAC-Man model.
* Participated in a field survey.

Exclusion criteria:

* Decline informed consent.

The criteria for Focus Group Discussions is as follows:

Inclusion criteria:

* Age 18 years or older.
* MOH or implementing partner professional or lay health worker at a study site (such as nurses, community health workers, health surveillance assistants, and HIV diagnostic assistants)
* Generally familiar with the PAC-Man model and/or EMTCT/ EID service delivery at their site.

Exclusion criteria:

* Decline informed consent.

The criteria for Key Informant Interviews is as follows:

Inclusion criteria:

* Age 18 years or older.
* HIV/ EMTCT policy maker OR MOH/ PEPFAR implementing partner senior manager.
* Generally familiar with HIV and/or EMTCT/ EID service delivery.

Exclusion criteria:

* Decline informed consent.

The criteria for Implementation Actor Questionnaires is as follows:

Inclusion criteria:

* Age 18 years or older.
* Professional or lay health provider at a study site.
* Generally familiar with HIV and/or EMTCT/ EID service delivery at their site.
* Participated in a focus group discussion.

Exclusion criteria:

* Decline informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2426 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants who receive EID testing by age 6 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants exposed to HIV who receive EID testing by age 6 months among the enumerated cohort of MIPs with infants at least 6 weeks old at all study sites.

SECONDARY OUTCOMES:
Proportion of infants who receive EID testing by age 2 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants exposed to HIV who receive EID testing by age 2 months among the enumerated cohort of all MIPs with infants at least 6 weeks old at all study sites.
Proportion of infants who receive EID testing by age 12 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants exposed to HIV who receive EID testing by age 12 months among the enumerated cohort of all MIPs with infants at least 6 weeks old at all study sites.
Proportion of high-risk infants who receive EID testing by age 6 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants with high-risk mothers exposed to HIV who receive EID testing by age 6 months among all high-risk MIPs with infants at least 6 weeks old at all study sites.
Proportion of infants who initiate ART | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants newly diagnosed with HIV who initiate ART ≤60 days from EID sample collection among the enumerated cohort of all infants.
Median infant results return time | Within 12 months of MIP enrollment in the national EMTCT program
  Median number of days from infant EID sample collection to results returned to caregivers.
Proportion of infants newly diagnosed with HIV | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants newly diagnosed with HIV among the enumerated cohort of all infants.
Median age at ART initiation among infants | Within 12 months of MIP enrollment in the national EMTCT program
  Median age in months at ART initiation among infants who test positive for HIV.
Median time to ART initiation among infants | Within 12 months of MIP enrollment in the national EMTCT program
  Median number of days to ART initiation among infants who test positive for HIV.
Proportion of infants who initiate ART the same day as diagnosis | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants newly diagnosed with HIV who initiate ART on the same day as EID results received among the enumerated cohort of all infants.
Proportion of infants with HIV retained in care at 3 months post-ART initiation | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants with HIV who are retained in care at 3-months post-ART initiation.
Proportion of infants with HIV retained in care at 6 months post-ART initiation | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of infants with HIV who are retained in care at 6-months post-ART initiation.
Proportion of MIPs reached with viral load testing | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of mothers living with HIV who received MOH-recommended 6-monthly VL testing during pregnancy and breastfeeding among the enumerated cohort of all MIPs.
Proportion of high-risk MIPs reached with viral load testing | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of high-risk MIPs living with HIV who received MOH-recommended 6-monthly VL testing during pregnancy and breastfeeding among all high-risk MIPs from the enumerated cohort.
Proportion of MIPs virally suppressed at 6 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of mothers with viral suppression (<1,000 copies of HIV per ml.) at 6 months after EMTCT enrollment among the enumerated cohort of all MIPs.
Proportion of high-risk MIPs virally suppressed at 6 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of high-risk mothers with viral suppression (<1,000 copies of HIV per ml.) at 6 months after EMTCT enrollment among the enumerated cohort of all MIPs.
Proportion of MIPs virally suppressed at 12 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of mothers with viral suppression (<1,000 copies of HIV per ml.) at 12 months after EMTCT enrollment among the enumerated cohort of all MIPs.
Proportion of high-risk MIPs virally suppressed at 12 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of high-risk mothers with viral suppression (<1,000 copies of HIV per ml.) at 12 months after EMTCT enrollment among the enumerated cohort of all MIPs.
Proportion of MIPs retained in care at 6 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of mothers who are retained in care (≥1 clinic encounter within the last 180 days) at 6 months after EMTCT enrollment among the enumerated cohort of all MIPs.
Proportion of MIPs retained in care at 12 months | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of mothers who are retained in care (≥1 clinic encounter within the last 180 days) at 12 months after EMTCT enrollment among the enumerated cohort of all MIPs.
Proportion of MIPs who resumed ART | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of mothers who had documented treatment interruption (i.e., a treatment gap ≥28 days) who later resumed ART among the enumerated cohort of all MIPs.
Proportion of MIPs who received enhanced adherence counseling | Within 12 months of MIP enrollment in the national EMTCT program
  Proportion of MIPs who had unsuppressed viral load and then completed enhanced adherence counselling among the enumerated cohort of all MIPs.
Adoption - proportion of sites that adopt the PAC-Man model | 6-12 months after sites switch to intervention; study endline (Approximately 12 months from the time that last study sites are switched to the intervention)
  Number of trained sites that deliver the PAC-Man intervention divided by the total number of trained sites. Study endline sustainability survey is conducted at the end of the trial once all study sites have been randomized to receive the intervention.
Adoption - proportion of providers who adopt the PAC-Man model | 6-12 months after sites switch to intervention; study endline (Approximately 12 months from the time that last study sites are switched to the intervention)
  Number of trained providers who deliver the PAC-Man intervention divided by the total number of trained providers. Study endline sustainability survey is conducted at the end of the trial once all study sites have been randomized to receive the intervention.
Implementation - cost per pediatric case | 6-12 months after sites switch to intervention; study endline (Approximately 12 months from the time that last study sites are switched to the intervention)
  Incremental cost of PAC-Man implementation per pediatric HIV case identified, compared to standard of care. Study endline sustainability survey is conducted at the end of the trial once all study sites have been randomized to receive the intervention.
Implementation - cost per unsuppressed MIP | 6-12 months after sites switch to intervention; study endline (Approximately 12 months from the time that last study sites are switched to the intervention)
  Incremental cost of PAC-Man implementation per pregnant and breastfeeding woman with unsuppressed viral load identified, compared to standard of care. Study endline sustainability survey is conducted at the end of the trial once all study sites have been randomized to receive the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herce, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- Malawi (3):
  - Bwaila Hospital, Lilongwe, Central Region
  - Area 18 Health Centre, Lilongwe
  - Monkey Bay Community Hospital, Monkey Bay

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with The University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Herce ME, Cassidy C, Munson A, Edwards JK, Rutstein SE, Matoga M, Kumwenda C, Simon KR, van Oosterhout JJ, Cox CM, Kamanga F, Kumwenda W, Phiri S, Rambiki E, Thawani A, Huwa J, Malewezi B, Mvalo T, Bula A, Chinula L, Hoffman I, Squibb MA, Nyirenda RK, Saidi F, Hosseinipour MC, Chagomerana MB. Study design and procedures for a hybrid effectiveness-implementation incomplete stepped-wedge cluster-randomized trial to evaluate a differentiated point-of-care HIV diagnosis and management model for the prevention of vertical transmission of HIV in Malawi: The PAC-Man trial protocol. Implement Sci Commun. 2025 Jul 28;6(1):78. doi: 10.1186/s43058-025-00762-5. PMID 40721832